CLINICAL TRIAL: NCT05905601
Title: User-centered Design of a Mobile Health Intervention to Promote Help-seeking and Reduce Duration of Untreated Illness Among Young Adults With Early Psychosis
Brief Title: mHealth for Psychosis Help-seeking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Buck, Assistant Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00009039; K23MH122504-01 (NIH)
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Psychosis
Keywords: Early psychosis; Psychosis risk; Duration of untreated psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NORTH "Full" (Experimental): Participants in the experimental arm will be provided access to the "Full" NORTH smartphone application designed to support young adults at risk for psychosis. They will also have access to the research team by phone for technical troubleshooting and support as necessary.
  Interventions: Behavioral: NORTH "Full"
- NORTH "Lite" (Experimental): Participants in the control arm will be provided access to the NORTH "Lite" smartphone application designed to support young adults at risk for psychosis. They will also have access to the research team by phone for technical troubleshooting and support as necessary.
  Interventions: Behavioral: NORTH "Lite"

INTERVENTIONS:
Behavioral: NORTH "Full" — NORTH is a native mobile app that provides on-demand content to young adults at risk for psychosis to improve or maintain their well-being, coping skills, and healthy habits, knowledge of psychosis, and provide help-seeking resources.
  Arms: NORTH "Full"
Behavioral: NORTH "Lite" — NORTH "Lite" contains the same on-demand lessons, practices and tracking features found in the "Full" NORTH mobile application but does not include help-seeking resources.
  Arms: NORTH "Lite"

SUMMARY:
The proposed study research project aims to develop and test a mobile health intervention designed to improve the wellness of young people at risk for psychosis and facilitate users' engagement with treatment and thus reduce duration of untreated psychosis. This clinical trial will involve a remote pilot randomized controlled trial that will examine (1) the feasibility of the proposed research approach, (2) the acceptability and usability of the NORTH intervention as well as (3) the specific additive value of help-seeking support in the context of self-guided mHealth for early psychosis. The full intervention, which includes psychoeducational lessons, Cognitive-Behavior Therapy-based practices, a symptom tracking feature, and help-seeking resources will be compared to a "Lite" version that will include the lessons, practices, and tracking but exclude the help-seeking resources.

ELIGIBILITY:
Inclusion Criteria:

* Elevated risk for psychosis that warrants further evaluation (a distress score >= 20 on the Prodromal Questionnaire, Brief [PQ-B], per Savill et al., 2018; and a positive frequency average score >= 1.47 on the Community Assessment of Psychic Experiences [CAPE-P15], per Jaya et al., 2021 and Bukenaite et al., 2017) and confirmation of symptoms consistent with online data collection checks (per Moritz et al., 2013)
* Age 18-30 years old
* Lives in the United States
* Under five years since participant's first psychotic episode or awareness of symptom onset
* Owns an iPhone
* Unengaged in specialty mental health treatment, in which the participant has not done either of the following in the previous three months: (1) taken a prescribed antipsychotic medication, (2) attended regular (i.e. more than one session of) psychotherapy.

Exclusion Criteria:

* Failed to demonstrate understanding of study details in comprehension screening process.
* Engaged in specialty mental health treatment in the previous three months, defined as the following: (1) taken a prescribed antipsychotic medication, OR (2) attended regular (i.e. more than one session of) psychotherapy.
* Unengaged in treatment, but only as a result of having completed or "graduated" from a specialty mental health program.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Buck, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NORTH "Full": Participants in the experimental arm will be provided access to the "Full" NORTH smartphone application designed to support young adults at risk for psychosis. They will also have access to the research team by phone for technical troubleshooting and support as necessary.
  NORTH: NORTH is a native mobile app that provides on-demand content to young adults at risk for psychosis to improve or maintain their well-being, coping skills, and healthy habits, knowledge of psychosis, and provide help-seeking resources.
Period: Overall Study
Arm/Group | NORTH "Full" | NORTH "Lite"
Started | 30 | 30
Completed | 29 | 27
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NORTH "Full" | NORTH "Lite" | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.20 (3.94) | 22.23 (3.82) | 22.22 (3.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 27 | 23 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 10 | 14
  White | 14 | 14 | 28
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Treatment Seeking Steps
Description: Treatment seeking will be measured using the Measure to Assess Steps to Service (MASS). The MASS is a 17-item self-report assessment of steps taken towards the attainment of mental health treatment, including research, social support, and engagement with service provider steps. Each item is endorsed on a three-point Likert scale (0 = No, I have not done this, 1 = I have done this once or twice, 2 = I have done this multiple times). The MASS is scored by summing individual items with higher scores indicating greater levels of treatment-seeking actions (range from 0 to 34). Increases in MASS scores were intended as an outcome of the proposed study (i.e. encouraging help-seeking).
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 6.43 (4.69) | 10.08 (7.08)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 7.65 (5.18) | 9.58 (7.33)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 8.17 (6.71) | 9.49 (8.09)

2. Primary Outcome: Change in Treatment-related Attitudes/Beliefs (Treatment Beliefs)
Description: Help-Seeking Attitudes and Stigma will be measured primarily using the Endorsed and Anticipated Stigma Inventory (EASI). The full EASI is a 40-item self-reported questionnaire with subscales measuring beliefs about mental illness, beliefs about mental health treatment, beliefs about mental health treatment seeking, concerns about stigma from loved ones, and concerns about stigma from the workplace. The subscales are scored by summing the ratings from the eight individual items in each subscale (5-point scale with 1 = Strongly disagree, 5 = Strongly agree), with lower scores indicating less stigma, and more positive attitudes towards treatment and treatment-seeking.
  The Beliefs About Treatment Scale assesses individuals' beliefs about the efficacy and usefulness of mental health treatments. It is totaled as a sum, and thus scores range from 8 to 40 with higher scores indicating more stigmatizing attitudes toward treatment.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 20.16 (4.87) | 18.47 (5.43)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 19.14 (4.82) | 19.13 (4.90)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 18.95 (5.24) | 17.78 (6.55)

3. Primary Outcome: Change in Treatment-related Attitudes/Beliefs (Treatment Seeking Attitudes)
Description: Help-Seeking Attitudes and Stigma will be measured primarily using the Endorsed and Anticipated Stigma Inventory (EASI). The full EASI is a 40-item self-reported questionnaire with subscales measuring beliefs about mental illness, beliefs about mental health treatment, beliefs about mental health treatment seeking, concerns about stigma from loved ones, and concerns about stigma from the workplace. The subscales are scored by summing the ratings from the eight individual items in each subscale (5-point scale with 1 = Strongly disagree, 5 = Strongly agree), with lower scores indicating less stigma, and more positive attitudes towards treatment and treatment-seeking.
  The Beliefs About Treatment Seeking assesses individuals' attitudes toward seeking mental health treatments. It is totaled as a sum, and thus scores range from 8 to 40 with higher scores indicating more stigmatizing attitudes toward treatment seeking.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 22.47 (4.87) | 21.50 (5.71)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 22.17 (6.08) | 22.44 (7.70)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 21.55 (6.12) | 21.26 (8.51)

4. Primary Outcome: Change in Internalized Stigma
Description: The Internalized Stigma of Mental Health Inventory, Brief (ISMI-9) will provide additional insight into the strength of participants' internalized stigma of mental illness. The ISMI-9 is a nine-item self-report short form, where each item is rated on a four-point Likert scale (1 = Strongly disagree, 4 = Strongly agree), and totaled as a mean score. Thus scores range from 1 to 4 with higher scores indicating more severe internalization of mental illness stigma.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants who completed fewer than half of the items on the scale are excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 2.34 (0.50) | 2.35 (0.40)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 2.29 (0.59) | 2.22 (0.59)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 2.26 (0.50) | 2.24 (0.58)

5. Primary Outcome: Change in Perceived Stress**
Description: Perceived stress will be measured using the Perceived Stress Questionnaire (PSQ), which is a 30-item, self-report questionnaire that examines the experience of stress independent of a specific and objective occasion. Items are endorsed on a four-point scale (1 = Almost never, 4 = Usually), and are summed for a total score (ranging from 30 to 120), with higher scores indicating higher levels of perceived stress.
  **NOTE: At baseline, the version provided to participants included the version of the PSQ that instructing participants to report on the past "year or two" while 6-week and 12-week assessments ask participants to report on the previous "month or so." While totals are still reported (as these still provide some information about intervention effects) these numbers should be interpreted with caution and in concert with other collected measures that include items about stress levels and coping with consistent reporting periods at all time points.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 87.14 (14.76) | 92.33 (12.52)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 82.97 (15.28) | 89.36 (12.13)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 79.66 (18.35) | 85.40 (14.70)

6. Primary Outcome: Change in Resilience / Coping
Description: The Brief Resilience Scale (BRS) will be used to assess resiliency. The BRS is a self-report form that consists of six resiliency statements that participants agree or disagree with on a five-point scale (1 = Strongly disagree, 5 = Strongly agree). Scores are totaled as a mean, and thus range from 1 to 5, with higher scores indicating greater resilience.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 2.69 (0.78) | 2.63 (0.95)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 2.70 (0.72) | 2.82 (1.01)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 2.74 (0.73) | 2.92 (1.04)

7. Secondary Outcome: Change in Symptoms (Positive)
Description: The Community Assessment of Psychic Experiences (CAPE-42) will be used to assess positive, negative and depressive symptoms of psychosis. The CAPE-42 is a self-report, 42 two-part item assessment that measures both the frequency of experiencing symptoms (four-point scale, 1 = Never, 4 = Almost Always) as well as the distress level (four-point scale, 1 = Not Distressed, 4 = Very Distressed) associated with each endorsed symptom. The CAPE weighted score can be calculated by summing the frequency and distress item responses. The positive subscale is 20 items and is totaled as a mean response ranging from 2 to 8, with higher scores indicating more frequent and distressing positive symptoms.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 3.44 (0.88) | 4.03 (1.05)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 3.42 (1.04) | 3.68 (1.15)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 3.18 (0.99) | 3.55 (1.15)

8. Secondary Outcome: Change in Symptoms (Negative)
Description: The Community Assessment of Psychic Experiences (CAPE-42) will be used to assess positive, negative and depressive symptoms of psychosis. The CAPE-42 is a self-report, 42 two-part item assessment that measures both the frequency of experiencing symptoms (four-point scale, 1 = Never, 4 = Almost Always) as well as the distress level (four-point scale, 1 = Not Distressed, 4 = Very Distressed) associated with each endorsed symptom. The CAPE weighted score can be calculated by summing the frequency and distress item responses. The negative subscale is 14 items and is totaled as a mean response ranging from 2 to 8, with higher scores indicating more frequent and distressing negative symptoms.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 4.54 (0.87) | 4.85 (1.33)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 4.39 (1.00) | 4.38 (1.10)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 4.35 (1.31) | 4.43 (1.22)

9. Secondary Outcome: Change in Symptoms (Depressive)
Description: The Community Assessment of Psychic Experiences (CAPE-42) will be used to assess positive, negative and depressive symptoms of psychosis. The CAPE-42 is a self-report, 42 two-part item assessment that measures both the frequency of experiencing symptoms (four-point scale, 1 = Never, 4 = Almost Always) as well as the distress level (four-point scale, 1 = Not Distressed, 4 = Very Distressed) associated with each endorsed symptom. The CAPE weighted score can be calculated by summing the frequency and distress item responses. The depressive subscale is 8 items and is totaled as a mean response ranging from 2 to 8, with higher scores indicating more frequent and distressing depressive symptoms.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 4.90 (1.20) | 5.32 (1.10)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 4.61 (1.28) | 4.61 (1.29)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 4.47 (1.40) | 4.75 (1.44)

10. Secondary Outcome: Change in Recovery
Description: Recovery will be assessed using the Choice of Outcome in CBT for Psychoses, Short Form (CHOICE-SF). The CHOICE-SF is an 11-item self-report form developed to assess recovery-related goals for therapy. Participants rate themselves in different therapy-focused areas such as "self-confidence" or "ways of dealing with everyday stress" on a scale (0 = Worst, 10 = Best). Scores on the CHOICE-SF are totaled as mean score across all standard items, and thus range from 0 to 10 with higher scores reflecting improved recovery.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 4.88 (1.42) | 4.77 (1.96)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 5.06 (1.52) | 5.23 (1.37)
  12 weeks: number analyzed (Participants) | 29 | 27
  12 weeks | 5.25 (1.59) | 5.54 (1.74)

11. Secondary Outcome: Change in Functioning
Description: Functioning will be measured using the Sheehan Disability Scale (SDS). The SDS is a short, five-item self-report form that assesses disability and functional impairment. The total score is the sum of three items measure to what extent symptoms have disrupted different aspects of daily life on a scale (0 = Not at all, 10 = Severely), thus the scale ranges from 0 to 30 with higher scores indicating greater functional impairment.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline: number analyzed (Participants) | 30 | 27
  Baseline | 16.27 (5.30) | 17.85 (6.90)
  6 weeks: number analyzed (Participants) | 29 | 27
  6 weeks | 14.21 (6.16) | 14.65 (7.64)
  12 weeks: number analyzed (Participants) | 27 | 27
  12 weeks | 12.76 (7.27) | 14.31 (7.57)

12. Secondary Outcome: Intervention Acceptability / Usability
Description: Usability/Acceptability will be assessed with a modified version of the System Usability Scale derived from our group's previous work developing mHealth interventions. This composite measure, which comprises 26 items based on four measures - the System Usability Scale, Post Study System Usability Scale, Technology Assessment Model Measurement Scales, and Usefulness, Satisfaction and Ease Questionnaire - assesses participants' experiences with the intervention during the study period (1 = Disagree, 2 = Neutral, 3 = Agree). While this measure is often interpreted qualitatively by item, we will also compare the overall score, which will comprise an average and thus range from 1 to 3, with higher scores reflecting higher acceptability and usability.
Time Frame: 6 weeks
Population: Participants are only analyzed if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NORTH "Full" | NORTH "Lite"
Number analyzed (Participants) | 29 | 27
score on a scale | 2.71 (0.20) | 2.71 (0.22)

ADVERSE EVENTS:
Time Frame: Full duration of study period, 3 months
Arm/Group | NORTH "Full" | NORTH "Lite"
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT05905601/Prot_SAP_000.pdf